CLINICAL TRIAL: NCT05297188
Title: The Effect of Ergonomic Sleep Mask Usage on Sleep Quality and Comfort in Intensive Care Patients
Brief Title: The Effect of Ergonomic Sleep Mask Usage on Patients' Sleep Quality and Comfort
Status: Completed | Type: Observational
Sponsor: Bartın Unıversity (Other)
Collaborators: Zonguldak Ataturk State Hospital (Other)
Responsible Party: Principal Investigator, Sevim Çelik, Professor Doctor, Bartın Unıversity
Other Study IDs: 2020-FEN-B-010
Record Dates: First submitted 2022-02-10; First posted 2022-03-28 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Sleep; Patient Compliance; Intensive Care Unit Acquired Weakness
Keywords: intensive care nursıng; surgıcal patient; sleep; ergonomic sleep mask
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- experimental group: Patients will be divided into experimental and control groups by block randomization. No application will be applied to the experimental group for first night sleep. On the morning of the first night, patients' comfort levels and sleep quality will be measured by Visual Analogue Scale and Richard-Campbell Sleep Scale. The second night, an ergonomic sleep mask will be worn to this group. In the morning of the second night, patients' comfort and sleep quality will be measured with the same scales. The patients will be asked to sleep between 22.00 and 24.00 on the second night, and intensive care lights will decrease, the noise level will be minimized, and patients will not wake up during the night outside their treatment.
  Interventions: Device: ergonomic sleep mask
- control group: Patients will be divided into experiment and control groups by block randomization. No application will be made to the control group for sleep on the first night. On the morning of the first night, patients' comfort levels and sleep quality will be measured by Visual Analogue Scale and Richard-Campbell Sleep Scale. On the second night, ear plugs and eye mask will be worn to this group. In the morning of the second night, patients' comfort and sleep quality will be measured with the same scales. Patients will be asked to sleep between 22.00 and 24.00 on the second night, and intensive care lights will decrease, noise level will be minimized and patients will not wake up during the night outside their treatment. It will be collected using the form.

INTERVENTIONS:
Device: ergonomic sleep mask — Ergonomic sleep mask; It is a material that covers the eye and ear completely and can be adjusted according to the patient, can be washed and reused at 30 degrees after use, 95% cotton, 5% polyester structure and 100% light proof properties.
  Groups: experimental group

SUMMARY:
In intensive care units, the sleep quality of patients decreases considerably due to reasons such as alarm sounds of some special devices, the number of healthcare professionals working in comparison to other clinics, their circulation is high, and the lights are constantly on.Studies conducted in intensive care units to facilitate the transition of patients to sleep and to improve sleep quality;has revealed that non-pharmacological applications increase sleep time and quality, reduce sleep disturbance,delirium,post-traumatic stress disorder and duration of stay in the intensive care unit.Although wearing earplugs and eye masks is a cost-effective and safe method and can improve perceived sleep quality in patients,eye masks and ear plugs are sometimes not comfortable.While the ear plugs dislocate during night sleep may cause the patients to wake up again,there are also situations such as the eye masks not being sized properly for the patients' eyes,and the part of the mask surrounding the head is thin and tense, disturbing the patient.By eliminating this situation that disturbs the patients, other solutions are needed to increase the quality of sleep without being affected by intensive care light and noise.

The project was planned to determine the effect of the ergonomic sleep mask on the sleep quality and comfort of patients in surgical patients whose treatment and care continues in intensive care units.The sample of the project consists of 128 patients by performing power analysis.Patients will be divided into two groups as 64 randomized patients in the control and experimental groups by applying block randomization.While there is no application to the experimental and control groups on the first night, an ergonomic sleep mask will be worn to the experimental group,and an ear plug and eye mask will be worn to the control group.At the end of the first night and the second night, the sleep quality of the patients will be evaluated with the 'Richard Campell Sleep Scale' and their comfort levels with the 'Visual Analogue Scale'.The data of the project will be collected using the Patient Information Form prepared in accordance with the literature. In the analysis of the data,Mann-Whitney U test, t test in independent groups, one-way ANOVA test and correlation analysis will be done.

DETAILED DESCRIPTION:
Human is an entity with physiological, biological, psychological, social and cultural needs. The basic needs required to sustain human life must be met. One of the basic needs to be met is 'sleep'. Sleep is a physiological requirement for people. Sleep, which makes up an average of 1/3 of human life; it is a process that causes changes in breathing, cardiac function, muscle tone, body temperature, hormone secretion and blood pressure. This process is the period of resting the body, repairing the cells, renewing the memory, arranging the memory functions and preparing for a new day.

Sleep status can be affected by many factors such as age, gender, diseases, environment, physical activity, nutrition, lifestyle, work life, medication, stimulant or smoking, and emotional state. Treatment and care processes related to patients undergoing surgical intervention also appear as one of the factors that significantly affect sleep. Surgical patients who are under threat before or after the surgery or who need special care because of the tools and equipment on the patient such as the drain and probe can remain in the intensive care unit for a while.

Intensive care units (ICUs) are the most dynamic, versatile and fast units circulating of hospitals where advanced technological tools and equipment are used to provide the highest level of benefit to life-threatened individuals, where highly educated physicians and nurses specializing in the care of critical patients are available. In the intensive care units, the sleep quality of patients due to the alarm sounds of some special devices, the work of health professionals more than other clinics, the circulation is high and the lights are constantly on decreases significantly. In the study conducted by Little et al., 116 intensive care patients were shown as the most common cause of sleep deprivation, 43% noise, 40% pain, 35% position impairment, 33% loud speech, 33% inserted catheters, and 29% time orientation disorder.Although the problem of insomnia in intensive care may vary according to studies, this rate is generally high. In the studies, it was stated that 75% of the patients experienced sleep problems due to noise, alarm sounds were the leading causes of noise, and the most obvious complaints of patients about sleep were waking up significantly.

For those patients who have problems such as pain, hunger, and discomfort from the foreign equipment (probe, drain, etc.) in their body after the surgery, insomnia causes their pain to feel more severe and decrease the comfort level. The use of more opioids to reduce the increasing pain, on the other hand, may cause the patients' recovery time to be extended as it will delay the important criteria such as early mobilization and early nutrition, which are important for the recovery of surgical patients. Therefore, patients should be provided to spend the night well. One of the main objectives of nursing care in intensive care units; to reduce the negative effects of the unit on the patient, to ensure the comfort of the patient, to reduce the anxiety of the patient and to facilitate the treatment by ensuring the patient's compliance with the ICU. Therefore, in order to reduce the existing pains of surgical patients, to be mobilized early, to switch to early nutrition, they should use the factors that help them to get enough sleep.

In intensive care units, non-pharmacological applications performed in order to facilitate the transition of patients to sleep and to improve sleep quality are superior to pharmacological applications with many advantages. Pharmacological applications should not be the first choice due to many reasons such as unnecessary drug use, side effects of drugs, drug interactions. Made studies revealed that non-pharmacological applications increase sleep time and quality, reduce sleep disturbance, delirium, post-traumatic stress disorder and duration of stay in the intensive care unit. In a large-scale systematic study, the effect of non-pharmacological applications on sleep quality was examined and although these applications had significant effects, the advantages and disadvantages of each application were mentioned separately.

As non-pharmacological methods to isolate patients from noise and light of intensive care units (ear plugs, eye mask etc.) the effects of single or combined use of equipment on patients' sleep quality have been discussed in many studies. In a study evaluated using the Pittsburgh Sleep Quality İndex, it was found that the quality of sleep significantly increased in the group using the eye mask. In another study conducted in the intensive care unit, eye mask and sleep plug were used together and it was revealed that there was a statistically significant difference between the delay in falling asleep, the quality of sleep and the length of sleep. It was found that the sleep quality in the experimental group significantly increased the Verran and Snyder-Halpern Sleep Scale subscales (discomfort, efficacy and supplement). In a study using the Richards Campbell Sleep Scale, the first test and posttest were applied to the experimental group and the control group, and the experimental group slept more hours after using eye mask and ear plugs, and a better perceived sleep quality was reported.

Although wearing earplugs and eye masks is a cost-effective and safe method and can improve perceived sleep quality in ICU patients, more research is needed to demonstrate the effect of this method. In addition, eye mask and ear plugs are sometimes not comfortable. While the ear plugs dislocate during night sleep may cause the patients to wake up again, the eye masks are not sized properly for the patients' eyes and if the thread surrounding the head of the masks is thin and tight, it may be disturbing the patient.

It is important that the eye mask and ear plugs are easier to use for the comfort of the patient and the material used can be adjusted according to the head and ear structure of the patient. For this reason, in the planned project, it was aimed to examine the effect of ergonomic sleep mask on 95% cotton, 5% polyester structure, which covers the eye and ear by covering it completely, adjustable according to the patient, can be washed and reused in a machine at 30 degrees after use.

ELIGIBILITY:
Inclusion Criteria:

* Acceptance for treat and care of intensive care unit following surgery
* Inpatient stay in the first 24 hours
* Volunteering to participate in the research
* Being 18 years of age or older
* Being able to communicate (patients with a minimum of Glaskow Coma Scale score of 12)
* Stable vital signs (arterial blood pressure, heart rate, oxygen saturation, body temperature)

Exclusion Criteria:

* No surgical intervention
* The length of stay in the intensive care unit after the surgery is not on the first day
* Having head, neck, ear and eye surgery
* Having eye and ear infections
* Chronic sleep disorder experience
* Sedation
* Having an allergy
* Depending on invasive or noninvasive mechanical ventilation
* Using assistive hearing aids
* Finding vision loss
* No communication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of the study, treatment and care in the intensive care unit of a public hospital attached to the Ministry of Health in Turkey consist of all patients who sustain. The sample group; after surgery, admitted to the intensive care unit and hospitalized within the first 24 hours, volunteering to participate in the study, communicable with patients 18 years of age and older (with a minimum of 12 GCS score), stable vital signs (arterial blood pressure, heartbeat rate, oxygen saturation, body temperature) will be created from patients. According to the literature review, the sample size was calculated as 128 using the G-POWER program with 0.5 effect size, 80% power and 0.5 error margin. Randomization will be made in the experimental and control groups, 64 patients each.
Sampling Method: Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
To compare the effects of using ergonomic sleep mask and ear plugs and eye mask on the comfort levels of patients in intensive care unit. | 1 year
  The effects on the comfort levels of the patients will be measured with the Visual Analog Scale.
  Visual Analog Scale: Using a ruler, the score is determined by mea-suring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. Based on the distribution of pain VAS scores in post- surgical patients (knee replacement, hyster-ectomy, or laparoscopic myomectomy) who described their postoperative pain intensity as none, mild, moderate, or severe, the following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm) (11). Normative values are not available. The scale has to be shown to the patient otherwise it is an auditory scale not a visual one.
To compare the effects of using ergonomic sleep mask and ear plugs and eye mask on sleep quality of patients in intensive care unit. | 1 year
  The effects on the sleep quality of the patients will be measured with the Richard-Campbell Sleep Scale.
  Richard-Campbell Sleep Scale: Developed by Richards in 1987, the RCSQ is a 6-item scale that evaluates the depth of night sleep, the time it takes to fall asleep, the frequency of awakening, the time to stay awake when awakened, the quality of sleep, and the noise level in the environment. Each item is evaluated on a chart between 0 and 100 using the visual analog scale technique. A score of "0-25" from the scale indicates very bad sleep, and a score of "76-100" indicates very good sleep. The total score of the scale is evaluated over 5 items, and the 6th item, which evaluates the noise level in the environment, is excluded from the total score evaluation. As the score of the scale increases, the sleep quality of the patients also increases. The Cronbach α value of the scale developed by Richards was found to be 0.82.

SECONDARY OUTCOMES:
To examine the effects of the type of anesthesia applied during the surgery on comfort of the patients staying in the intensive care units after surgery. | 1 year
  The effects on comfort of the patients will be measured with the Visual Analog Scale.
  Visual Analog Scale: Using a ruler, the score is determined by mea-suring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. Based on the distribution of pain VAS scores in post- surgical patients (knee replacement, hyster-ectomy, or laparoscopic myomectomy) who described their postoperative pain intensity as none, mild, moderate, or severe, the following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm) (11). Normative values are not available. The scale has to be shown to the patient otherwise it is an auditory scale not a visual one.
To examine the effects of the type of anesthesia applied during the surgery on sleep quality of the patients staying in the intensive care units after surgery. | 1 year
  The effects on sleep quality of the patients will be measured with the Richard-Campbell Sleep Scale.
  Richard-Campbell Sleep Scale: Developed by Richards in 1987, the RCSQ is a 6-item scale that evaluates the depth of night sleep, the time it takes to fall asleep, the frequency of awakening, the time to stay awake when awakened, the quality of sleep, and the noise level in the environment. Each item is evaluated on a chart between 0 and 100 using the visual analog scale technique. A score of "0-25" from the scale indicates very bad sleep, and a score of "76-100" indicates very good sleep. The total score of the scale is evaluated over 5 items, and the 6th item, which evaluates the noise level in the environment, is excluded from the total score evaluation. As the score of the scale increases, the sleep quality of the patients also increases. The Cronbach α value of the scale developed by Richards was found to be 0.82.
To examine the effects of the type of surgery applied to patients on the sleep quality of patients staying in the intensive care units after surgery. | 1 year
  The effects on the sleep quality of the patients will be measured with the Richard-Campbell Sleep Scale.
  Richard-Campbell Sleep Scale: Developed by Richards in 1987, the RCSQ is a 6-item scale that evaluates the depth of night sleep, the time it takes to fall asleep, the frequency of awakening, the time to stay awake when awakened, the quality of sleep, and the noise level in the environment. Each item is evaluated on a chart between 0 and 100 using the visual analog scale technique. A score of "0-25" from the scale indicates very bad sleep, and a score of "76-100" indicates very good sleep. The total score of the scale is evaluated over 5 items, and the 6th item, which evaluates the noise level in the environment, is excluded from the total score evaluation. As the score of the scale increases, the sleep quality of the patients also increases. The Cronbach α value of the scale developed by Richards was found to be 0.82.
To examine the relationship between the socio-demographic characteristics of patients and their comfort status in the intensive care units. | 1 year
  The effects on the comfort of the patients will be measured with the Visual Analog Scale.
  Visual Analog Scale: Using a ruler, the score is determined by mea-suring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. Based on the distribution of pain VAS scores in post- surgical patients (knee replacement, hyster-ectomy, or laparoscopic myomectomy) who described their postoperative pain intensity as none, mild, moderate, or severe, the following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm) (11). Normative values are not available. The scale has to be shown to the patient otherwise it is an auditory scale not a visual one.
To examine the relationship between the socio-demographic characteristics of patients and their sleep quality in the intensive care units. | 1 year
  The effects on the comfort of the patients will be measured with the Richard-Campbell Sleep Scale.
  Richard-Campbell Sleep Scale: Developed by Richards in 1987, the RCSQ is a 6-item scale that evaluates the depth of night sleep, the time it takes to fall asleep, the frequency of awakening, the time to stay awake when awakened, the quality of sleep, and the noise level in the environment. Each item is evaluated on a chart between 0 and 100 using the visual analog scale technique. A score of "0-25" from the scale indicates very bad sleep, and a score of "76-100" indicates very good sleep. The total score of the scale is evaluated over 5 items, and the 6th item, which evaluates the noise level in the environment, is excluded from the total score evaluation. As the score of the scale increases, the sleep quality of the patients also increases. The Cronbach α value of the scale developed by Richards was found to be 0.82.
To examine the relationship between the patients' intensive care experiences and their sleep quality after the night they spent in the intensive care unit. | 1 year
  The effects on the sleep quality of the patients will be measured with the Richard-Campbell Sleep Scale.
  Richard-Campbell Sleep Scale: Developed by Richards in 1987, the RCSQ is a 6-item scale that evaluates the depth of night sleep, the time it takes to fall asleep, the frequency of awakening, the time to stay awake when awakened, the quality of sleep, and the noise level in the environment. Each item is evaluated on a chart between 0 and 100 using the visual analog scale technique. A score of "0-25" from the scale indicates very bad sleep, and a score of "76-100" indicates very good sleep. The total score of the scale is evaluated over 5 items, and the 6th item, which evaluates the noise level in the environment, is excluded from the total score evaluation. As the score of the scale increases, the sleep quality of the patients also increases. The Cronbach α value of the scale developed by Richards was found to be 0.82.
To examine the relationship between the patients' intensive care experiences on comfort after the night they spent in the intensive care unit. | 1 year
  The effects on comfort of the patients will be measured with the Visual Analog Scale.
  Visual Analog Scale: Using a ruler, the score is determined by mea-suring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. Based on the distribution of pain VAS scores in post- surgical patients (knee replacement, hyster-ectomy, or laparoscopic myomectomy) who described their postoperative pain intensity as none, mild, moderate, or severe, the following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm) (11). Normative values are not available. The scale has to be shown to the patient otherwise it is an auditory scale not a visual one.

CONTACTS AND LOCATIONS:
Locations (1):
- Bartın University, Merkez, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No